CLINICAL TRIAL: NCT05355792
Title: Clinical Investigation Title: An Open, Prospective, Multicenter Investigation to Evaluate the Clinical Outcome of OmniTaper EV Implants in Extraction Sockets and Healed Ridges - A 5-year Follow-up
Brief Title: Multicenter Study to Evaluate the Clinical Outcome of the OmniTaper EV Implant in Single Tooth Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-OM-21-002
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Jaw, Edentulous
Keywords: Partially
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single tooth restorations (Experimental): A single, open-label group with patients in need of single tooth restorations will receive an OmniTaper EV implant system available in the following sizes: diameter 3.4, 3.8, 4.5 and 5.5 mm and lengths 8, 9.5, 11, 13, 15 and 18 mm.
  Interventions: Device: OmniTaper EV implants

INTERVENTIONS:
Device: OmniTaper EV implants — Partially edentulous subjects in need of one implant in the maxilla or mandible (2nd and 3rd molars excluded) will receive an OmniTaper EV implant system. The study will be done in accordance with standard dental practice using a one- or two-stage surgical protocol and immediate or delayed placement and/or loading.
  Other Names: OmniTaper EV implants UDI 0739253224012WR

SUMMARY:
This clinical study, funded by the company Dentsply Sirona, is being carried out to see if the newly developed tooth implant "OmniTaper EV" is safe, effective and functions as intended when replacing a lost or removed tooth. The OmniTaper EV implant is a further development of existing dental implants. It is made of titanium, a metal that is well tolerated by the human body, which has been successfully used in dental implants for more than 40 years. All components used in this study are available on the market, are CE-marked and will be used according to intended use and approved instructions.

The study involves at 11 planned clinic visits including follow-up visits 6 months and annually until 5 years after installation of the permanent crown. after over a period of about five and a half years. The treatment method and healing period may vary depending on the individual case and treatment plan and additional visits may therefore need to be scheduled. The visits and procedures are the same as standard of care and no procedures will be done just for purpose of research.

The study aims to recruit about 137 men and women from six clinics across Europe (Germany, UK and Switzerland) and participants can only receive one study implant each. Participation is entirely voluntary and participants can choose to withdraw from the study at any time, without giving a reason. The decision to decline or withdraw participation will not affect participants future treatment or care

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign and date the informed consent form.
* In need of an implant in position 16 to 26 or 36 to 46 (2nd and 3rd molars are excluded), and each subject can only receive one implant.
* Deemed by the PI/Subinvestigator as likely to present with an initially stable implant situation.
* A stable occlusion, i.e. an opposing natural dentition, a crown, an implant-supported fixed or removable prosthesis, a partial removable prosthesis or a full denture.
* An adjacent tooth (root with natural or artificial crown) or an implant-supported crown mesially and distally. Exemption: If the planned implant is in the first molar position, an edentulous space is accepted distally

Exclusion Criteria:

* Not willing to participate in the clinical investigation or not able to understand the content of the clinical investigation.
* Unlikely to be able to comply with clinical investigation procedures according to PI's/Subinvestigator's judgement.
* Unable or unwilling to return for follow-up visits for a period of 5 years.
* Severe non-compliance to CIP as judged by the PI/Subinvestigator and/or Dentsply Sirona.
* Known allergy or hypersensitivity to titanium and/or stainless steel.
* Uncontrolled pathological process in the oral cavity, e.g. untreated rampant caries and uncontrolled periodontal disease.
* Uncontrolled para-functional habits, e.g. bruxism.
* Current need of any Guided Bone Regeneration (GBR) procedure in the planned implant area (gap filling at immediate placement and soft tissue grafting are allowed).
* Systemic or local disease or condition that would compromise post-operative healing and/ or osseointegration.
* Immunosuppression, use of corticosteroids, prior or current use of oral or intravenous bisphosphonate, or any other medication such as anti-resorptive therapy or monoclonal antibodies that could compromise post-operative healing and/or osseointegration.
* Any other condition that would make the subject unsuitable for participation, including but not limited to:

  * History of radiation therapy in the head and neck region.
  * History of chemotherapy within 5 years prior to surgery.
  * Present alcohol and/or drug abuse.
  * Ongoing psychiatric illness.
  * Current smoking/use of tobacco, including e-cigarettes /Not applicable for UK).
* Any ongoing disease that would make the subject unsuitable for participation, including but not limited to:

  * Recent myocardial infarction (< 3 months*).
  * Recent cerebrovascular accident (< 3 months*).
  * Recent cardiac-valvular prosthesis placement (< 3 months*).
  * Hemorrhagic diathesis.
  * Severe liver dysfunction.
  * Known or suspected current malignancy.
  * Uncontrolled diabetes mellitus (as reported by the subject).
  * Florid infection.
* Pregnant or breastfeeding females. (Pregnancy tests will be performed as per local requirements).
* Previous enrolment in the present clinical investigation.
* Involvement in the planning and conduct of the clinical investigation (applies to both Dentsply Sirona personnel and the clinical investigation site).
* Simultaneous participation in another clinical investigation, or participation in a clinical investigation during the last 6 months that may interfere with the present clinical investigation.

'* < 3 months is a strict exclusion criterion. After 3 month it is up to the investigator to judge whether the subject is considered suitable for participation or not.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate 1 year after permanent restoration by counting implant in place 1 year after permanent restoration | 1 year after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Implant survival rate is a binary variable evaluated clinically, i.e. 'Yes' or 'No' where 'Yes' means that the implant is still in place and 'No' means that the implant is not in place. Any implant that has been removed or lost after implant placement visit will be considered a failure, whatever the reason for removal/loss.

SECONDARY OUTCOMES:
Implant survival rate at 3 and 5 years after permanent restoration by counting implant in place. | 3 and 5 year after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Implant survival rate is a binary variable evaluated clinically, i.e. 'Yes' or 'No' where 'Yes' means that the implant is still in place and 'No' means that the implant is not in place. Any implant that has been removed or lost after implant placement visit will be considered a failure, whatever the reason for removal/loss.
Change of implant stability quotient value (ISQ) between implant placement and permanent restoration. | From date of implant placement (which is estimated to occur approximately 1 month after enrollment).
  Implant stability will be evaluated by ISQ value using Resonance Frequency Analysis (RFA). The stability is presented as an ISQ value. The higher the ISQ value the higher the stability. Recorded as a numeric value (1-100).
Final and maximum insertion torque value for each implant at implant placement. | At date of implant placement (which is estimated to occur approximately 1 month after enrollment).
  Final and maximum insertion torque value (ITV), based on ITV curve, measured in Ncm.
Surgeon's assessment of implant stability and confidence at implant placement for each implant. | Immediately after implant placement (which is estimated to occur approximately 1 month after enrollment).
  Numerical scale 1-10, where 1 = totally disagree with the statement, and 10 = totally agree with the statement. Statements to be evaluated by the surgeon: "The implant was guided into the prepared osteotomy", "The implant followed the prepared osteotomy", "The implant has a good primary stability". Each statement will be evaluated separately.
Implant success, i.e., number of implants documented as successful at 1, 3 and 5 years after permanent restoration. | 1, 2, 3 and 5 years after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Successful implants counted, i.e. 'Yes' or 'No'. An implant will be considered successful if all of the following criteria are fulfilled:
  Implant in place. Lack of evidence of peri-implant radiolucency in X-ray. Less than 1mm vertical bone loss during first year after loading with permanent restoration and 0,2mm annually thereafter.
  Absence of persistent and/or irreversible signs and symptoms such as pain, infections, neuropathies, paresthesia, or violation of the mandibular canal.
Maintenance of marginal bone levels (MBL). | At permanent restoration (which is estimated to occur approximately 3 months after implant placement) and at 1, 3 and 5 years after PR..
  The MBL change from permanent restoration compared to 1, 3, and 5 years. MBLs will be determined from X-rays, expressed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant. The average will be calculated and compared for each evaluation period.
PPD (Probing Pocket Depth) | At PR (which is estimated to occur approximately 3 months after implant placement) and at 1, 2, 3, 4 and 5 years after PR.
  PPD will be evaluated at four surfaces around the implant (mesial, distal, buccal and lingual), by using a periodontal probe. The distance from the mucosal margin to the bottom of the probe-able pocket will be measured in millimeter. PPD mean values will be calculated on an implant level for each visit. Changes over time will be analyzed.
Bleeding on Probing (BoP) | At PR (which is estimated to occur approximately 3 months after implant placement) and at 1, 2, 3, 4 and 5 years after PR.
  BoP will be evaluated at four surfaces around the implant (mesial, distal, buccal and lingual), by using a periodontal probe. Bleeding will be recorded as presence or absence of bleeding when probing to the bottom of the pocket. The proportion of surfaces with presence of bleeding will be calculated and presented on an implant level for each visit.
Plaque | 6 months, 1, 2, 3, 4 and 5 years after PR (which is estimated to occur approximately 3 months after implant placement).
  Plaque will be recorded as presence or absence of plaque by visual inspection on four surfaces at each implant site.The proportion of surfaces with presence of plaque will be calculated and presented on an implant level for each visit.
Occurrence of Adverse Events (AEs) | From date of implant placement (which is estimated to occur approximately 1 month after enrollment) up to 5 years after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Continuously collected and reported AEs at each investigation visit from implant placement.
Occurrence of Adverse Device Effects (ADEs) | From date of implant placement (which is estimated to occur approximately 1 month after enrollment) up to 5 years after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Continuously collected and reported ADEs at each investigation visit from implant placement.
Occurrence of Device Deficiencies (DDs) | From date of implant placement (which is estimated to occur approximately 1 month after enrollment) up to 5 years after permanent restoration (which is estimated to occur approximately 3 months after implant placement).
  Continuously collected and reported DDs at each investigation visit from implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gehrke, Dr, Principal Investigator — Praxis Prof. Dr. Dhom & Kollegen MVZ GmbH Bismarckstraße, Ludwigshafen, Germany
Locations (6):
- Germany (3):
  - Praxis Prof. Dr. Dhom & Kollegen MVZ GmbH, Ludwigshafen
  - Private Clinic Schloss Schellenstein, Olsberg
  - Kornmann Gerlach & Kollegen, Oppenheim
- Dr. med. dent. Alessandro Hellmuth Ponte, Lugano, Switzerland
- United Kingdom (2):
  - The Implant Experts, Maidstone, Kent
  - Birmingham Dental Hospital, Birmingham, West Midlands